CLINICAL TRIAL: NCT04227951
Title: A Randomised Multicentre Controlled Trial of Gastrectomy With or Without Prophylactic Abdominal Drainage. The Abdominal Drain in Gastrectomy Trial (ADiGe Trial)
Brief Title: Gastrectomy With or Without Drainage (ADiGe)?
Acronym: ADiGe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2245CESC
Record Dates: First submitted 2020-01-08; First posted 2020-01-14 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer
Keywords: Gastrectomy; Drain; Drainage
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Masking Description: The leading surgeon and the patient will be blinded to the arm assigned until the end of the operation. No blinding is provided for the patient, care providers, or coordinating researcher after the operation. After the operation we thought that was unreliable to go ahead with participants blindness considering that one arm has an evident drain and the other arm has no drain. Considering that clinicians will need to check drain quality and remove the tube in treatment group we considered not possible to mask the care providers or investigators on this practice.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain (Sham Comparator): Participants enrolled in this arm have an abdominal drain positioned at the end of the operation (any type, inserted from right flank with the tip close to the esophago-jejunal or Gastro-jejunal anastomosis and the duodenal stump). Drain will stay in place until postoperative day (POD) 4th (drain output and quality will be registered). If normal drain debt and patient have no abdominal complications that need reoperation and/or percutaneous drain placement until POD 4, a methylene-blue test is be performed (200 ml water + 5 ml blue orally, check drain after 60 minutes: negative test if no blu was seen in the drain). If negative-blue test drain can be removed according to centre preference (no strict POD defined); if positive-blue test complication will be treated according to centre preference. Only in this arm drain related complications are registered. Need for reoperation and/or percutaneous drain placement (primary outcome) are registered.
  Interventions: Device: Drain placement
- No Drain (Experimental): Participants enrolled in this arm do not have any abdominal drain placed at the end of the operation. Postoperative management (e.g. resume of oral intake, anastomosis integrity tests) is left to centre preference. Need for reoperation and/or percutaneous drain placement (primary outcome) are registered.
  Interventions: Device: Avoid drain placement

INTERVENTIONS:
Device: Avoid drain placement — In No Drain arm (experimental) no abdominal drain is placed at the end of the operation.
  Arms: No Drain
Device: Drain placement — In Drain arm (sham comparator) an abdominal drain is inserted in the abdomen from the right flank, passing below the liver (close to the duodenal stump) with the apex behind the esophago-jejunal (in total gastrectomy) or gastro-jejunal (in subtotal gastrectomy) anastomosis.
  Arms: Drain

SUMMARY:
Prophylactic use of anastomotic drain in upper gastrointestinal surgery has been questioned in the last 15 years but only small studies have been conducted. In 2015 a Cochrane meta analysis on four Randomized Controlled Trials (RCT) concluded that there was no convincing evidence to the routine drain placement in gastrectomy. Nevertheless the Authors evidenced the moderate/low methodological quality of the included studies and highlighted how 3 out of four came from Eastern countries. Despite the above mentioned limits, Enhanced Recovery After Surgery (ERAS) society published the guidelines for gastrectomy that strongly recommend, with high evidence level, to avoid routine use of drain in gastric surgery. After 2015 some other retrospective studies have been published, all with inconsistent results. Our objective is to perform a multicentre prospective trial in a large western cohort of patients to establish wether avoid routine use of anastomotic drain does not led to an increasing of postoperative invasive procedure.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients that undergo total or subtotal gastrectomy with a curative intent, for histologically proven gastric cancer or esophago-gastric junction cancer Siewert type II or III, in surgical investigator centres from the beginning of the study until reaching the accrual number
* esophageal involvement <= 2 cm
* patients undergoing upfront surgery or treated with a neoadjuvant/perioperative chemotherapy
* open, hybrid, laparoscopic or robotic approach
* all types of anastomosis (circular stapled, linear stapled, hand sewn)

Exclusion Criteria:

* refuse to sign informed consent
* age <18
* Heart failure New York Heart Association (NYHA) class IV
* severe liver disease (Child >= 7)
* pregnancy
* metastatic disease
* emergency surgery
* palliative surgery
* operation different from total or subtotal oncological gastrectomies (e.g. pylorus preserving, proximal gastrectomy)
* lymphnodal dissection <D1
* reconstruction different from Roux-en-Y or Billroth II
* multiple organ resections (except for cholecystectomy)
* gastric cancer with duodenal involvement
* intraoperative Hyperthermic Intraperitoneal Chemotherapy (HIPEC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
30 day reoperation AND/OR additional drain placement | 30 days after the operation
  Incidence of reoperation AND/OR percutaneous placement of an additional drain within postoperative day 30 (composite outcome)

SECONDARY OUTCOMES:
Overall mortality | 90 days after the operation
Overall morbidity | 30 days after the operation OR in hospital if hospitalization is longer than 30 days, up to 90 days of hospitalization
  Complications are classified according to International consensus on a complications list after gastrectomy for cancer - Baiocchi et Al, Gastric Cancer, 2019 and stratified according to Clavien-Dindo classification.
Length of hospital stay | From the day of operation until discharge (home or other facilities) or death for any cause whichever came first, assessed up to 100 months.
Drain related complications | From the day of operation until drain removal up to 90 days after the operation
  Only in Drain Group complications related to drain placement (e.g. bleeding from drain site) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni de Manzoni, Prof, Principal Investigator — Università degli studi di Verona
Locations (11):
- Italy (11):
  - Ospedale Morgagni di Forlì - Chirurgia generale, Forlì, Forlì-Cesena
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga- Chirurgia Generale, Orbassano, Torino
  - Policlinico San Marco, GSD - Chirurgia Generale ed Oncologica, Bergamo
  - Policlinico S.Orsola-Malpighi - Dipartimento di Chirurgia Generale, Bologna
  - Ospedale di Cremona, Cremona
  - Ospedale San Raffaele - Chirurgia Gastroenterologica -, Milan
  - ASST Grande Ospedale metropolitano Niguarda - Chirurgia generale oncologica e mini-invasiva, Milan
  - Azienda Ospedaliero Universitaria Modena - Chirurgia Oncologica, Generale e d'Urgenza, Modena
  - Ospedale Federico II di Napoli- Chirurgia Generale, Napoli
  - Azienda Ospedaliera Universitaria Parma - UO Clinica Chirurgica Generale, Parma
  - Azienda Ospedaliera Universitaria Integrata Borgo Trento - Chirurgia Generale ed Esofago Stomaco, Verona

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in abdominal surgery. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact jacopo.weindelmayer@aovr.veneto.it

REFERENCES:
- [Background] Wang Z, Chen J, Su K, Dong Z. Abdominal drainage versus no drainage post-gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2015 May 11;2015(5):CD008788. doi: 10.1002/14651858.CD008788.pub3. PMID 25961741
- [Background] Mortensen K, Nilsson M, Slim K, Schafer M, Mariette C, Braga M, Carli F, Demartines N, Griffin SM, Lassen K; Enhanced Recovery After Surgery (ERAS(R)) Group. Consensus guidelines for enhanced recovery after gastrectomy: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Br J Surg. 2014 Sep;101(10):1209-29. doi: 10.1002/bjs.9582. Epub 2014 Jul 21. PMID 25047143
- [Background] Schots JPM, Luyer MDP, Nieuwenhuijzen GAP. Abdominal Drainage and Amylase Measurement for Detection of Leakage After Gastrectomy for Gastric Cancer. J Gastrointest Surg. 2018 Jul;22(7):1163-1170. doi: 10.1007/s11605-018-3789-7. Epub 2018 May 7. PMID 29736661
- [Background] Dann GC, Squires MH 3rd, Postlewait LM, Kooby DA, Poultsides GA, Weber SM, Bloomston M, Fields RC, Pawlik TM, Votanopoulos KI, Schmidt CR, Ejaz A, Acher AW, Worhunsky DJ, Saunders N, Swords DS, Jin LX, Cho CS, Winslow ER, Russell MC, Staley CA, Maithel SK, Cardona K. Value of Peritoneal Drain Placement After Total Gastrectomy for Gastric Adenocarcinoma: A Multi-institutional Analysis from the US Gastric Cancer Collaborative. Ann Surg Oncol. 2015 Dec;22 Suppl 3:S888-97. doi: 10.1245/s10434-015-4636-7. Epub 2015 May 29. PMID 26023037
- [Background] Hirahara N, Matsubara T, Hayashi H, Takai K, Fujii Y, Tajima Y. Significance of prophylactic intra-abdominal drain placement after laparoscopic distal gastrectomy for gastric cancer. World J Surg Oncol. 2015 May 12;13:181. doi: 10.1186/s12957-015-0591-9. PMID 25962503
- [Background] Lee J, Choi YY, An JY, Seo SH, Kim DW, Seo YB, Nakagawa M, Li S, Cheong JH, Hyung WJ, Noh SH. Do All Patients Require Prophylactic Drainage After Gastrectomy for Gastric Cancer? The Experience of a High-Volume Center. Ann Surg Oncol. 2015 Nov;22(12):3929-37. doi: 10.1245/s10434-015-4521-4. Epub 2015 Apr 7. PMID 25845430
- [Derived] Weindelmayer J, Mengardo V, Ascari F, Baiocchi GL, Casadei R, De Palma GD, De Pascale S, Elmore U, Ferrari GC, Framarini M, Gelmini R, Gualtierotti M, Marchesi F, Milone M, Puca L, Reddavid R, Rosati R, Solaini L, Torroni L, Totaro L, Veltri A, Verlato G, de Manzoni G; Italian Research Group for Gastric Cancer (GIRCG). Prophylactic Drain Placement and Postoperative Invasive Procedures After Gastrectomy: The Abdominal Drain After Gastrectomy (ADIGE) Randomized Clinical Trial. JAMA Surg. 2025 Feb 1;160(2):135-143. doi: 10.1001/jamasurg.2024.5227. PMID 39602143
- [Derived] Weindelmayer J, Mengardo V, Veltri A, Baiocchi GL, Giacopuzzi S, Verlato G, de Manzoni G; Italian Research Group for Gastric Cancer (GIRCG). Utility of Abdominal Drain in Gastrectomy (ADiGe) Trial: study protocol for a multicenter non-inferiority randomized trial. Trials. 2021 Feb 17;22(1):152. doi: 10.1186/s13063-021-05102-1. PMID 33596959